CLINICAL TRIAL: NCT01213472
Title: Study of GSK2241658A Antigen-Specific Cancer Immunotherapeutic in Patients With Unresectable and Progressive Metastatic Cutaneous Melanoma
Brief Title: Evaluation of a New Anti-cancer Immunotherapy in Patients With Non-operable and Progressing Metastatic Cutaneous Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112406; 2010-020663-20 (EudraCT Number)
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Melanoma
Keywords: ASCI; melanoma; tumor antigen; unresectable; progressive; NY-ESO-1; adult; cancer-testis antigen; Immunotherapy
MeSH Terms: conditions — Melanoma

ARMS (1):
- NY-ESO 1 Group (Experimental): Patients with non-operable and progressing metastatic cutaneous melanoma, received up to 24 doses of GSK2241658A Cancer Immunotherapeutic, provided that at each tumor evaluation time point, the clinical criteria to continue the treatment were met, including patients having a clinical response.
  Interventions: Biological: GSK Biologicals' 2241658A Antigen-Specific Cancer Immunotherapeutic (ASCI)

INTERVENTIONS:
Biological: GSK Biologicals' 2241658A Antigen-Specific Cancer Immunotherapeutic (ASCI) — Up to 24 intramuscular administrations

SUMMARY:
The purpose of this study is to investigate the safety, immunogenicity and clinical activity of GSK2241658A antigen-specific cancer immunotherapeutic (ASCI) for the treatment of patients with non-operable and progressing metastatic cutaneous melanoma.

DETAILED DESCRIPTION:
In this study, patients were to receive a maximum of 24 doses of recNY-ESO-1 + AS15 ASCI according four cycles over a period of four years. An active follow-phase (up to five years after registration into the study) was planned for all patients.

As of Amendment 3, there will no longer be an active follow-up of patients after discontinuation or completion of the treatment. The study will end 30 days after the last dose will be administered.

In addition, no more biological samples will be collected for protocol research purposes. For each biological sample already collected in the scope of this study and not tested yet, testing will not be performed by default, except if a scientific rationale remains relevant.

Blood sampling for safety monitoring as per protocol will continue.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient with histologically proven, measurable metastatic cutaneous melanoma, and with documented progressive disease within the 12 weeks before the first administration of study treatment.
* Written informed consent for NY-ESO-1 expression screening and gene profiling on resected tumor tissue and for the complete study has been obtained from the patient prior to shipment of the sample for expression testing and prior to the performance of any other protocol-specific procedure.
* Patient is >= 18 years of age at the time of signature of the informed consent.
* The patient's tumor shows expression of NY-ESO-1, as determined by real-time quantitative reverse transcription polymerase chain reaction (RT-PCR) analysis or any updated technique on fresh tissue sample(s).
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* The patient has normal organ functions as shown by all of the following:

  * Hemoglobin ≥ 12 g/dL
  * Absolute leukocytes count ≥ 3.0 x 1000000000/L
  * Absolute lymphocytes count ≥ 1.0 x 1000000000/L
  * Platelets ≥ 100 x 1000000000/L
  * Serum creatinine ≤ Upper Limit of Normal (ULN)
  * Serum total bilirubin ≤ 1.5 x ULN (except for patients with Gilbert's syndrome for whom the limit is 2 x ULN)
  * Lactate dehydrogenase ≤ ULN
  * Aspartate aminotransferase ≤ 2 × ULN
  * Alanine aminotransferase ≤ 2 × ULN

These tests must be done no more than 3 weeks before the first ASCI administration.

* Female patients of non-childbearing potential may be enrolled in the study.
* Female patient of childbearing potential may be enrolled in the study, if the patient:

  * has practiced adequate contraception for 30 days prior to first ASCI administration, and
  * has a negative pregnancy test at the specified study visits, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the ASCI administration series.
* In the view of the investigator, the patient can and will comply with the requirements of this protocol.

Exclusion Criteria:

* The patient has at any time received systemic chemotherapy, biochemotherapy, small molecules or nti-CTLA-4 monoclonal antibody for metastatic disease.
* The patient is scheduled to receive any other anticancer treatments than those specified in the protocol, including but not limited to (bio-) chemotherapeutic, immunomodulating agents and radiotherapy.
* The patient received any cancer immunotherapy containing a NY-ESO-1 antigen or any cancer immunotherapy for his/her metastatic disease.
* The patient requires concomitant treatment with systemic corticosteroids, or any other immunosuppressive agents.
* Use of any investigational or non-registered product other than the ASCI within 30 days preceding the first ASCI administration, or planned use during the study period.
* The patient has (had) previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers or carcinoma in situ of the cervix or effectively treated malignancy that has been in remission for over 5 years and is highly likely to have been cured.
* The patient has an allergy to any component of the study investigational product or has a history of previous allergic reactions to vaccinations.
* The patient has an autoimmune disease such as, but not limited to, multiple sclerosis, lupus, and inflammatory bowel disease. Patients with vitiligo are not excluded.
* The patient has a family history of congenital or hereditary immunodeficiency.
* The patient is known to be positive for the Human Immunodeficiency Virus.
* The patient has an uncontrolled bleeding disorder.
* The patient has a family history of congenital or hereditary immunodeficiency.
* The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent, or to comply with the trial procedures.
* The patient has concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
* For female patients: the patient is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-01-31 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- Australia (2):
  - GSK Investigational Site, North Sydney, New South Wales
  - GSK Investigational Site, Woolloongabba, Queensland
- GSK Investigational Site, Graz, Austria
- France (4):
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
- Germany (4):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
- Italy (3):
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Siena, Tuscany
- Netherlands (3):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Rotterdam
- Switzerland (2):
  - GSK Investigational Site, Geneva
  - GSK Investigational Site, Zurich
- United Kingdom (3):
  - GSK Investigational Site, Chelmsford
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] American Joint Committee on Cancer. 2002. Cancer staging manual. Sixth edition. Springer editions.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Among 169 subjects screened, 33 were vaccinated and 6 completed the study. Following the NCT00480025 and NCT00796445 studies, which failed to demonstrate clinical efficacy of the MAGE-A3 antigen-specific cancer immunotherapeutic (ASCI), GSK decided to stop the development of ASCI studies and recruitment in ongoing studies.
Pre-assignment Details: Accordingly, patients still on treatment in the study, at the time of protocol amendment 3, either continued until last dose or until recurrence, whichever came first, or until patient or investigator decided to stop study treatment. Therefore, the results summary contain limited primary and secondary endpoints results, and are merely descriptive.
Period: Overall Study
Arm/Group | NY-ESO 1 Group
Started | 33
Completed | 6
Not Completed | 27
Not completed — Recurrence/Progressive disease | 25
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.7 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian / European Heritage | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Severe Toxicities During the Study Treatment Period
Description: Severe toxicity was defined, according to the Common Terminology Criteria for Adverse Events (CTCAE) (version 4.0), as 1)an Antigen-Specific Cancer Immunotherapeutic (ASCI) related or possibly related Grade 3 or higher toxicity. Grade 3 myalgia, arthralgia, headache, fever, rigors/chills and fatigue (including lethargy, malaise and asthenia) should persist for 48 hours despite therapy to be taken into account and as 2)an ASCI related or possibly related Grade 2 or higher allergic reaction occurring within 24 hours of the dose administration.
Time Frame: During the study treatment period (maximum duration = 49 months).
Population: The analysis was performed on the total treated cohort (TTC), which included all subjects who received at least one dose of the Antigen-Specific Cancer Immunotherapeutic (ASCI) treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 33
Participants | 0

2. Primary Outcome: Number of Patients With Severe Toxicities During the Follow-up Period
Description: Severe toxicity was defined, according to the Common Terminology Criteria for Adverse Events (CTCAE) (version 4.0), as 1)an Antigen-Specific Cancer Immunotherapeutic (ASCI) related or possibly related Grade 3 or higher toxicity. Grade 3 myalgia, arthralgia, headache, fever, rigors/chills and fatigue (including lethargy, malaise and asthenia) should persist for 48 hours despite therapy in order to be taken into account and as 2)an ASCI related or possibly related Grade 2 or higher allergic reaction occurring within 24 hours of the dose administration. All active follow-up visits and procedures were stopped, hence this follow-up analysis was not performed as initially planned.
Time Frame: During the one year follow-up period (i.e. from Month 49 until Month 61)
Population: The analysis was to be performed on the total treated cohort (TTC), which included all subjects who received at least one dose of the ASCI treatment. All active follow-up visits and procedures were stopped, hence this follow-up analysis was not performed as initially planned.
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Patients With the Best Overall Response in the Overall Population
Description: Best response was recorded from the start of treatment until disease progression. Response assessment was essentially based on a set of measurable lesions (target lesions [TL]), and any other lesions (non-target lesions [NTL]), both identified at baseline. Complete Response (CR)=disappearance of all TL or NTL; Partial Response (PR) = at least 30 percent (%) decrease in the sum of the longest diameter(LD) of TL compared to baseline, stable disease (SD) = neither sufficient shrinkage to qualify PR nor sufficient increase to qualify for Progressive disease (PD) compared with baseline; PD = at least 20% increase in the sum of LD of TL compared with baseline, or the appearance of one or more new lesions, or both of these, and/or unequivocal progression of existing NTL; NE =non-evaluable; Clinical response: any CR or PR best overall response; Disease control: any CR, PR, SD or SD/PR best overall response.
Time Frame: During the study treatment period (maximum duration = 49 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 33
Participants
  Best response, CR | 3
  Best response, PR | 2
  Best response, SD | 2
  Best response, SD/PR | 2
  Best response, PD | 23
  Best response, NE | 1
  Clinical Response, Yes | 5
  Clinical Response, No | 28
  Disease control, Yes | 9
  Disease control, No | 24

4. Secondary Outcome: Number of Patients With Best Overall Response Including Mixed Response (MxR) and Slow Progressive Disease (SPD) Criteria
Description: Patients with Slow Progressive Disease (SPD) status met the following criteria: patient's Eastern Cooperative Oncology Group (ECOG) performance status was 0 or 1, patient's lactate dehydrogenase (LDH) value was not greater than twice the normal upper limit, there was no appearance of visceral metastases other than in the lung, patients did not meet any of the criteria for permanent stopping of study treatment. Mixed response (MxR) criteria was defined as follows: at least 30% decrease in the longest diameter (LD) occurring in at least one target lesion recorded and measured at baseline. Such response occurring in otherwise stable disease (SD) or progressive disease (PD) status of LD of target lesions and without the appearance of one or more new lesions were classified as "SD with target lesion regression" or "PD with target lesion regression". The appearance of new lesions in otherwise partial response (PR) status of the LD of target lesions were classified as "PR with new lesion".
Time Frame: During the study treatment period (maximum duration = 49 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 33
Participants
  CR | 3
  PR | 2
  SD/PR | 2
  MxR: SD with target lesion regression | 0
  MxR: PD with target lesion regression | 3
  MxR: PR with new lesion | 2
  SD without mixed response | 2
  PD with SPD criteria | 10
  PD without SPD/MxR | 8
  NE | 1

5. Secondary Outcome: Number of Patients With Objective Clinical Response (CR or PR) in the Population of Patients Who Present the Predictive Melanoma Antigen A3 (MAGE-A3) Gene Signature
Description: Following MAGE3-AS15-NSC-003 (ADJ) (NCT00480025) study (A double-blind, randomized, placebo-controlled Phase III study to assess the efficacy of recMAGE-A3 + AS15 Antigen-Specific Cancer immunotherapeutic as adjuvant therapy in patients with resected MAGE-A3-positive Non-Small Cell Lung Cancer) showed the absence of treatment effect in any of the primary, secondary, or exploratory analyses, clinical activity was not reported within the population of patients who present the predictive MAGE-A3 gene signature, in that study.
Time Frame: After 12, 22, 31 and 54 weeks of treatment.
Population: As study development was stopped earlier and decision was taken not to perform further testing on biological samples already collected, except if a scientific rationale remained relevant, analyses for patients who presented MAGE-A3 gene signature as required in this outcome, were not performed.
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Patients With Adverse Events (AEs) by Maximum Grade
Description: An AE is any untoward medical occurrence in a clinical investigation patient, temporally associated with the use of a medical product, whether or not considered related to the medicinal product. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e. lack efficacy), abuse or misuse.
Time Frame: During the study treatment period (maximum duration = 49 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 33
Participants
  Any event, Grade 1 | 9
  Any event, Grade 2 | 21
  Any event, Grade 3 | 3
  Any event, Grade 4 | 0
  Any event, Grade 5 | 0

7. Secondary Outcome: Number of Patients With Adverse Events (AEs) That Are Causally Related to Treatment Administration by Maximum Grade
Description: as for outcome 6
Time Frame: During the study treatment period (maximum duration = 49 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 33
Participants
  Any event, Grade 1 | 20
  Any event, Grade 2 | 13
  Any event, Grade 3 | 0
  Any event, Grade 4 | 0
  Any event, Grade 5 | 0

8. Secondary Outcome: Number of Patients With Serious Adverse Events (SAEs) by Maximum Grade
Description: A serious adverse event (SAE) is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study patient, is a grade 4 AE according to the Common Terminology Criteria for Adverse Events (CTCAE, v 4.0), in addition, in this study, Grade 3 or higher pIMDs were considered as medically significant and were therefore notified as SAE.
Time Frame: During the study treatment period (maximum duration = 49 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 33
Participants
  Any event, Grade 1 | 0
  Any event, Grade 2 | 1
  Any event, Grade 3 | 2
  Any event, Grade 4 | 0
  Any event, Grade 5 | 0

9. Secondary Outcome: Number of Patients With Serious Adverse Events (SAEs) That Are Causally Related to Treatment Administration by Maximum Grade
Description: A serious adverse event (SAE) is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study patient, is a grade 4 AE according to the Common Terminology Criteria for Adverse Events (CTCAE, v 4.0), in addition, in this study, Grade 3 or higher pIMDs will be considered as medically significant and will therefore be notified as SAE. No serious adverse events were reported during the study period that are causally related to treatment administration by maximum grade.
Time Frame: During the study treatment period (maximum duration = 49 months).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 33
Participants | 0

10. Secondary Outcome: Time to Treatment Failure (TTF)
Description: Time to Treatment Failure (TTF) was defined as the time from first treatment until the date of the last treatment administration, for patients who discontinued the treatment prematurely, regardless of the reason for study treatment discontinuation. Patients who completed their full treatment phase or who were still on treatment at the time of analysis were censored on their last study treatment administration date..
Time Frame: From first treatment administration (i.e. at Week 0) until the last treatment administration (i.e. at Month 48)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 33
Months | 4.7 [3.3 to 11.7]

11. Secondary Outcome: Progression-free Survival (PFS) Rate
Description: Progression-free survival (PFS) was defined as the time from first treatment to either the date of first disease progression (PD) or the date of death (for whatever reason), whichever came first. Patients alive and without disease progression were censored at the date of the last visit/contact.
Time Frame: From first treatment administration (i.e. at Week 0) until the last tumor evaluation (i.e. at Month 49)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 33
Months | 2.8 [2.8 to 2.9]

12. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from first treatment until death. Patients alive at the time of analysis were censored at the time of last visit/contact.
Time Frame: From first treatment administration (i.e. at Week 0) until the last tumor evaluation (i.e. at Month 49)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 33
Months | NA [NA to NA] — The median was not reached at the time of the analysis.

13. Secondary Outcome: The Duration of Response for Patients With CR, PR or Stable Disease (SD) Status
Description: The duration of response was measured from the time when the measurement criteria for CR/PR (whichever was recorded first) or SD evaluation were met until the first date that first PD or death was objectively documented (taking as reference for PD the smallest measurements recorded since the treatment started). Stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the sum of LD of target lesions recorded previously but not necessarily at baseline (The minimal time interval required between two measurements for determination of SD was at least 16 weeks.). The analysis was not performed as initially planned.
Time Frame: From first treatment administration (i.e. at Week 0) until the last tumor evaluation (i.e. at Month 49)
Population: As study development was stopped earlier and decision was taken not to perform further testing on biological samples already collected, except if a scientific rationale remained relevant, analyses on Duration of Response for Patients With CR, PR or SD Status, as required in this outcome, were not performed.
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Patients With Progression-free Survival Events
Description: Progression-free survival was defined as the time from the date of registration of the patient to either the date of disease progression or the date of death (for whatever reason), whichever came first. Patients alive and without disease progression were censored at the date of their last tumor evaluation. PFS events included progressive disease (PD), death in absence of PD and events (Any event which was part of the natural course of the disease under study, was captured as an efficacy measure. Therefore it did not need to be reported as an SAE).
Time Frame: From first treatment administration (i.e. at Week 0) until the last tumor evaluation (i.e. at Month 49)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 33
Participants
  PD, Yes | 29
  PD, No | 4
  Death in absence of PD, Yes | 0
  Death in absence of PD, No | 33
  Events, Yes | 29
  Events, No | 4

15. Secondary Outcome: Summary of Deaths Related to Progressive Disease of Cancer Under Study Reported After the Study Treatment, in the Period of Long-term Follow-up for Survival
Description: Summary of deaths included death, autopsy performed and cause of death. Progression of the tumor was recorded in the clinical assessments. Death due to progressive disease was to be recorded on a specific form in the case report form but not as a serious adverse event (SAE). However, if the investigator considered that there was a causal relationship between the administration of the treatment or protocol design/procedures and the disease progression, then this must be reported as an SAE.
Time Frame: During the long-term Follow-Up period for progressive disease and survival [1 year after the study treatment end (at Month 49) or up to 5 years after the first study treatment administration, regardless of disease progression and study discontinuation.]
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 33
Participants
  Death, Yes | 8
  Death, No | 25
  Autopsy performed, Yes | 0
  Autopsy performed, No | 6
  Autopsy performed, Unknown | 2
  Cause of death, Disease under study (melanoma) | 8

16. Secondary Outcome: Anti NY-ESO-1 Antibody Concentrations
Description: Anti-NY-ESO-1 antibody concentrations were presented as geometric mean concentrations (GMTs) and expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: Before treatment (PRE), at 4 (W4), 8 (W8), 10 (W10), 12 (W12), 29 (W29), 51 (W51), 75 (W75), 99 (W99), 123 (W123) weeks of treatment and at the concluding visit, i.e. at Month 49 (POST)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 27
EL.U/mL
  PRE | 179.7 [100.8 to 320.3]
  W4: number analyzed (Participants) | 26
  W4 | 4134.0 [2250.9 to 7592.3]
  W8: number analyzed (Participants) | 21
  W8 | 15235.4 [9762.1 to 23777.2]
  W10: number analyzed (Participants) | 23
  W10 | 22373.0 [15198.4 to 32934.5]
  W12: number analyzed (Participants) | 19
  W12 | 25626.1 [16866.9 to 38934.0]
  W29: number analyzed (Participants) | 13
  W29 | 30684.5 [22913.5 to 41091.2]
  W51: number analyzed (Participants) | 6
  W51 | 23393.6 [16574.2 to 33018.9]
  W75: number analyzed (Participants) | 4
  W75 | 12661.4 [8063.2 to 19881.9]
  W99: number analyzed (Participants) | 3
  W99 | 10313.6 [3389.6 to 31381.9]
  W123: number analyzed (Participants) | 2
  W123 | 5878.2 [1460.4 to 23659.5]
  POST: number analyzed (Participants) | 9
  POST | 17775.8 [10390.0 to 30411.8]

17. Secondary Outcome: Humoral Response for Anti NY-ESO-1 Antibodies
Description: Anti NY-ESO-1 antibody response was defined as: For initially seronegative patients: post-vaccination antibody concentration greater than or equal to (≥) 179 EU/mL and for intially seropositive patients: post-vaccination antibody concentration ≥ 2 fold the pre-vaccination antibody concentration.
Time Frame: At 4 (W4), 8 (W8), 10 (W10), 12 (W12), 29 (W29), 51 (W51), 75 (W75), 99 (W99), 123 (W123) weeks of treatment and at the concluding visit, i.e. at Month 49 (POST)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 26
Participants
  W4 | 24
  W8: number analyzed (Participants) | 21
  W8 | 21
  W10: number analyzed (Participants) | 23
  W10 | 23
  W12: number analyzed (Participants) | 19
  W12 | 19
  W29: number analyzed (Participants) | 13
  W29 | 13
  W51: number analyzed (Participants) | 6
  W51 | 6
  W75: number analyzed (Participants) | 4
  W75 | 3
  W99: number analyzed (Participants) | 3
  W99 | 1
  W123: number analyzed (Participants) | 2
  W123 | 0
  POST: number analyzed (Participants) | 9
  POST | 9

18. Secondary Outcome: Cell Mediated Immune Response for Anti-NY-ESO-1 Antibodies (T-cell)
Description: Cellular (T-cell) response was not analysed as data only available for few patients.
Time Frame: as for outcome 16
Population: As study development was stopped earlier, and decision was taken not to perform further testing on biological samples already collected, except if a scientific rationale remained relevant, Cellular (T-cell) response was not analysed as data only available for few patients.
Arm/Group | NY-ESO 1 Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected during the study treatment period, i.e. from Month 0 to Month 49 (maximum treatment duration) in the overall population. All-Cause Mortality events were collected during the long-term Follow-Up period for progressive disease and survival [1 year after the study treatment end (at Month 49) or up to 5 years after the first study treatment administration, regardless of disease progression and study discontinuation.]
Description: As planned per study protocol, any event which was part of the natural course of the disease under study was captured as an efficacy measure (i.e.: Progression of the tumor and death due to progressive disease) and did not need to be reported as an SAE or fatal SAE. However, if the investigator considered that there was a causal relationship between the administration of the ASCI or protocol design/procedures and the disease progression, then this was reported as an SAE.
Arm/Group | NY-ESO 1 Group
All-Cause Mortality (participants affected / at risk) | 8/33
Serious Adverse Events (participants affected / at risk) | 3/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NY-ESO 1 Group (N=33)
Anaemia (Blood and lymphatic system disorders) | 1
Postoperative wound infection (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Uterine cyst (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NY-ESO 1 Group (N=33)
Anaemia (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Periorbital oedema (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Oral pain (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Administration site rash (General disorders) | 1
Asthenia (General disorders) | 6
Chills (General disorders) | 5
Fatigue (General disorders) | 15
Impaired healing (General disorders) | 1
Inflammation (General disorders) | 1
Influenza like illness (General disorders) | 15
Injection site erythema (General disorders) | 6
Injection site induration (General disorders) | 2
Injection site inflammation (General disorders) | 1
Injection site oedema (General disorders) | 2
Injection site pain (General disorders) | 22
Injection site pruritus (General disorders) | 3
Injection site reaction (General disorders) | 6
Injection site swelling (General disorders) | 2
Malaise (General disorders) | 3
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 5
Pyrexia (General disorders) | 13
Swelling (General disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Bronchitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral viral infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 3
Tinea infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Bone contusion (Injury, poisoning and procedural complications) | 1
Graft complication (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Blood pressure decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Weight decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Tumor haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumor ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Disturbance in attention (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 11
Hypersomnia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 4
Neuropathy peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 3
Sciatica (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Irritability (Psychiatric disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Cervical polyp (Reproductive system and breast disorders) | 1
Uterine cyst (Reproductive system and breast disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 2
Hyperaemia (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Lymphoedema (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2014-09-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT01213472/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT01213472/SAP_001.pdf